CLINICAL TRIAL: NCT05111314
Title: Intraindividual Comparison of Hepatic Intraarterial Versus Systemic Intravenous 68Ga-PSMAPET/CT in Patients With HCC: Pilot Study
Brief Title: Comparison of Hepatic Intraarterial Versus Systemic Intravenous 68Ga-PSMA PET/CT for Detection of Hepatocellular Carcinoma
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI requested
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Scott M. Thompson, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 21-004930; NCI-2021-11290 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — gallium 68 PSMA-11; 68Ga-DKFZ-PSMA-11; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (embolization, 68Ga-PSMA, PET/CT) (Experimental): Patients undergoing clinically indicated hepatic artery embolization will receive 68Ga-PSMA intraarterially (IA) over 5 minutes. After 60-90 minutes, patients undergo PET/CT scan over 1 hour.
  Interventions: Radiation: Gallium Ga 68 Gozetotide; Procedure: Hepatic Artery Embolization; Procedure: Positron Emission Tomography and Computed Tomography Scan

INTERVENTIONS:
Radiation: Gallium Ga 68 Gozetotide — Given IA
  Other Names: (68)Ga labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; (68)Ga-labeled Glu-urea-Lys(Ahx)-HBED-CC; (68)Ga-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68)Gallium-PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; (68Ga)Glu-urea-Lys(Ahx)-HBED-CC; 68Ga-DKFZ-PSMA-11; 68Ga-HBED-CC-PSMA; 68Ga-labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; 68Ga-PSMA; 68Ga-PSMA-11; 68Ga-PSMA-HBED-CC; [68Ga] Prostate-specific Membrane Antigen 11; [68Ga]GaPSMA-11; Ga PSMA; Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled PSMA-11; GA-68 PSMA-11; Gallium Ga 68 PSMA-11; Gallium Ga 68-labeled PSMA-11; GALLIUM GA-68 GOZETOTIDE; Gallium-68 PSMA; Gallium-68 PSMA Ligand Glu-urea-Lys(Ahx)-HBED-CC; GaPSMA; PSMA-HBED-CC GA-68
Procedure: Hepatic Artery Embolization — Undergo hepatic artery embolization
Procedure: Positron Emission Tomography and Computed Tomography Scan — Undergo PET/CT scan
  Other Names: PET-CT Scan; PET/CT SCAN; Positron Emission Tomography/Computed Tomography

SUMMARY:
This phase 0/1 study evaluates intraarterial administration of gallium Ga 68 gozetotide (68Ga-PSMA) for the detection of prostate-specific membrane antigen (PSMA) positive liver cancer by positron emission tomography (PET)/computed tomography (CT). 68Ga-PSMA is an imaging agent used with PET/CT scans to locate PSMA positive lesions. This study evaluates intraarterial administration of this agent, compared to intravenous administration.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the tumor radiotracer uptake (first pass effect or regional advantage) of direct hepatic intraarterial (I.A.) versus systemic intravenous (I.V.) 68Ga-PSMA in patients with PSMA+ hepatocellular carcinoma (HCC) by PET/CT.

OUTLINE:

Patients undergoing clinically indicated hepatic artery embolization will receive 68Ga-PSMA intraarterially (IA) over 5 minutes. After 60-90 minutes, patients undergo PET/CT scan over 1 hour.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either an imaging diagnosis of HCC by CT or magnetic resonance imaging (MRI) (Liver Imaging and Reporting Data System 5 [LI-RADS 5]) confirmed by a board-certified abdominal radiologist, or with biopsy-proven HCC
* Already enrolled in ongoing Transform the Practice or Department of Defense 68Ga-PSMA studies
* PSMA avid HCC detected by 68Ga-PSMA PET/CT after intravenous administration of 68Ga-PSMA confirmed by a board certified nuclear radiologist
* Undergoing planned hepatic artery embolization (HAE) per standard clinical care
* Male or female with age greater than 18 years, with the capacity and willingness to provide a written informed consent

Exclusion Criteria:

* Subjects requiring emergent surgery for a ruptured/bleeding HCC
* Pregnant and/or breast-feeding subjects. A negative pregnancy test within 48 hours of the PET scan
* Subjects with higher than the weight/size limitations of PET/CT scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Intraindividual intralesional difference in maximum standardized uptake value (SUVmax) | Up to 2 years
  Intraindividual intralesional difference in maximum standardized uptake value (SUVmax) will be evaluated as fold change and absolute difference for a given lesion between intra-arterially (I.A.) and intravenous (I.V.) prostate-specific membrane antigen (PSMA) positron emission tomography (PET). Qualitative evaluation assesses the intensity of PSMA uptake in hepatic lesions, graded as follows: grade 1: uptake < normal liver; grade 2: uptake = normal liver; grade 3: uptake > normal liver; grade 4: uptake > spleen or kidneys. Semi-quantitative analysis is undertaken by calculating intraindividual difference in SUVmax for each lesion between I.A. and I.V. PSMA PET followed by a two-sided one sample t-test. Maximum and mean standardized uptake value (SUVmax, SUVmean, SUVmin) of the lesion(s), and SUVmax of the background liver are noted.

SECONDARY OUTCOMES:
Intraindividual intralesional differences in tumor to background (TBR) of SUVmax | Up to 2 years
  For each lesion, tumor-to-liver background ratio (TBR) of SUVmax will be calculated and the intraindividual intralesional difference in TBR of SUVmax will be compared on a lesion basis between I.A. and I.V. PSMA PET.
Difference in PSMA uptake measured by SUVmax (fold change, absolute difference) in the kidneys, spleen and salivary glands between I.A. and I.V. PSMA PET. | Up to 2 years
  SUVmax will be measured for the kidneys, spleen and salivary glands and the difference in PSMA uptake measured by SUVmax (fold change, absolute difference) in the kidneys, spleen and salivary glands will be compared between I.A. and I.V. PSMA PET
Incidence of adverse events | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott M Thompson, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States